CLINICAL TRIAL: NCT02940743
Title: Behavioral Management of Phosphorus in Hemodialysis
Brief Title: Behavioral Management of Phosphorus in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00817
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Disease (CKD); Hyperphosphatemia
Keywords: Hemodialysis
MeSH Terms: conditions — Cardiovascular Diseases; Hyperphosphatemia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education (Edu) (Active Comparator)
  Interventions: Behavioral: Education (Edu)
- Edu + Self-Monitoring (SM) (Active Comparator)
  Interventions: Behavioral: Education (Edu); Behavioral: SM intervention
- Edu + SM + Social Cognitive Theory (SCT) (Active Comparator)
  Interventions: Behavioral: Education (Edu); Behavioral: SM intervention; Behavioral: Social Cognitive Therapy (SCT)

INTERVENTIONS:
Behavioral: Education (Edu) — This intervention will take place during weeks 1-4 at the dialysis center. Each week, study staff will present participants with a brief educational video on: phosphorus binder adherence (week 1), meeting dietary protein needs (week 2), restricting dietary sources of phosphorus (week 3), and eliminating phosphorus-based food additives (week 4). These videos will be loaded onto tablet (Personal Computers) PCs so that participants can easily view them during regular dialysis treatment.
Behavioral: SM intervention — During the first 12 weeks of the intervention, a study dietitian will review the participants' records, and provide individualized feedback via a password-protected NYULMC email address. Feedback will be provided twice per week during weeks 1-4, once per week during weeks 5-8, and once every two weeks during weeks 9-12. The email messages will focus on both the importance of self-monitoring and the behavioral targets of the intervention. Feedback will use standardized language rather than specific dietary examples to avoid providing individualized counseling to participants (which is not the purpose of the SM intervention).
  Arms: Edu + SM + Social Cognitive Theory (SCT); Edu + Self-Monitoring (SM)
Behavioral: Social Cognitive Therapy (SCT) — This intervention will be delivered remotely online using the same tablet PCs provided for the SM intervention component of this treatment condition. The behavioral training program will focus on building a sense of self-efficacy with emphasis on mastery experiences that will include emphasizing past successes; setting incremental, easily achievable goals; self-monitoring to stay on track; identifying modifiable barriers to healthy behavior; positive feedback in goal achievement; and developing participant expertise in both the regimen and in problem solving around barriers to adherence.
  Arms: Edu + SM + Social Cognitive Theory (SCT)

SUMMARY:
The purpose of this randomized clinical trial is to evaluate alternative technology-supported behavioral approaches to engaging 42 maintenance hemodialysis (HD) patients with persistent hyperphosphatemia in phosphorus binder adherence and dietary phosphorus restriction. Participants will be randomized to 1 of 3 intervention groups: (1) Education (Edu); (2) Edu + Self-Monitoring (SM); or (3) Edu + SM + Social Cognitive Theory (SCT)-based training program.

DETAILED DESCRIPTION:
Investigators will evaluate the intervention in terms of feasibility and acceptability, behavior change at 12 and 24 weeks (reported phosphorus binder adherence, reported nutrient intakes, normalized protein catabolic rate), and clinical outcomes (serum phosphorus concentrations, symptoms). In addition, the impact of the different behavioral approaches on self-efficacy at 12 and 24 weeks, and the mediating effects of self-efficacy in facilitating behavioral changes and clinical outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Receiving thrice-weekly hemodialysis treatment for at least 3 months
* 3-month average serum phosphorus concentration >5.5 mg/dL

Exclusion Criteria:

* Unable to participate meaningfully in the combined Edu + SM + SCT intervention, including:
* Unable to read and/or speak English
* Self-monitoring application is currently available in English only (patients will not be excluded from participation on the basis of race/ethnicity)
* Cognitively-impaired
* Physically-impaired
* Institutionalized or otherwise having limited control over diet
* Life expectancy of <1 year per dialysis center staff
* Women who are pregnant or become pregnant during the study

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Hemodialysis (HD) patients that are eligible for the study | 24 Weeks
  Measure of feasibility
Proportion of eligible patients who agree to participate | 24 Weeks
  Measure of feasibility
Proportion of enrolled participants who complete the study | 24 Weeks
  Measure of Acceptability

SECONDARY OUTCOMES:
8-item Morisky Medication Adherence Survey (MMAS-8) | 24 Weeks
  Used to measure Binder Adherence, has been shown to be a valid and reliable measure of antihypertensive medication adherence
Reported dietary energy, protein and phosphorus intake | 2 Weeks
  participants will be directed to complete three, non-consecutive food records over the two-week period. Diet record days will include two weekdays (1 dialysis day and 1 non-dialysis day), and one non-dialysis weekend day.
Normalized protein catabolic rate (nPCR) | 24 Weeks
  The nPCR is an objective measure of protein intake in HD patients based on the accumulation of urea nitrogen in blood between dialysis treatments
Serum phosphorus. | 24 Weeks
  Pre-dialysis serum phosphorus concentrations are a key secondary clinical endpoint for this intervention. Serum phosphorus is already being measured in participants as part of the routine monthly laboratory blood work, so this information will be obtained from the participant's medical charts.
Frequency and severity of participant symptoms assessed via an investigator-developed questionnaire | 24 Weeks
  (itching, bone and joint pain, cramping) and phosphorus binders (difficulty defecating, loose or watery stools) will be self-reported via an investigator-developed questionnaire.
Balance Wise Self-Efficacy for Restricting Dietary Sodium in Hemodialysis Scale | 24 Weeks
  be adapted to focus on adherence to phosphorus binders, dietary phosphorus restrictions and adequacy of protein intake. The self-efficacy questionnaire asks participants' to report their confidence in the next month that they will be able to complete various tasked related to the study intervention. An overall scale, and subscale scores for phosphorus binders, dietary phosphorus restriction and adequacy of protein intake will be computed by summing pertinent items for analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sevick, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States